CLINICAL TRIAL: NCT07118852
Title: Developing Remote Human Milk Collection as a Novel Technique for Transcriptome Sequencing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-0663; Protocol Version 11/11/25 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison); Pending (Registry Identifier: ICTR award)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Human Milk
Keywords: sample collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Lactating Participants (Experimental)
  Interventions: Device: Remote Human Milk Sample Collection

INTERVENTIONS:
Device: Remote Human Milk Sample Collection — Two products will be evaluated for their ability to preserve RNA in human milk samples.
  * RNAlater (ThermoFisher©) (ratio variable)
  * NucleoProtect RNA (Takara©) (ratio variable)*
    * Product volume mixed with human milk samples will vary by product and may be titrated as part of protocol development.

SUMMARY:
This study will develop a protocol for remote human milk collection for use in gene expression research through application of ribonucleic acid (RNA) preservation reagents. The investigators hypothesize that addition of preservation reagents will preserve RNA in human milk, facilitating downstream analyses that require intact RNA. 50 lactating participants will be recruited and requested to provide reagent-mixed samples to be sent to the university through shipping services where they will be evaluated for RNA quantity, quality and profile.

DETAILED DESCRIPTION:
To preserve the quality of RNAs, commonly used methods for collecting fresh human milk samples typically require a stringent collection and handling routine. This includes proximity to a laboratory (within 20 minutes of driving distance) and ultra-cold storage conditions (below -80°C). Compared to "non-research" settings, current standards in sample collection require either 1) participant travel or 2) home visits for biospecimen collection. These requirements impede the inclusion of wide, non- biased milk samples from a range of populations, which is necessary for robust human subject studies. Subsequently, certain populations are excluded due to arbitrary factors like location, daytime availability, and residence. The development of human milk collection protocols that enable wide-ranging participation is a research priority that supports our research at the University of Wisconsin - Madison and any global investigative efforts that include human milk RNA sequencing.

Recruitment will take place in 2 phases (N=25 participants each) to allow for adjustments to the biospecimen collection kit and optimization of RNA integrity. During the first recruitment phase, N=25 participants will be recruited and enrolled using a reagent: human milk concentration of approximately 2:1.

After return of N=25 participant kits, recruitment will briefly pause to extract RNA and run RNA integrity analyses. Results of analyses will inform whether to proceed to phase 2 (recruitment and enrollment of an additional N=25 participants) with the same reagent: human milk concentrations or whether to adjust volume or concentration. Total volume of human milk collection will not exceed 30 mL.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and reading
* Lactating for greater than or equal to 4 weeks

Exclusion Criteria:

* not meeting personal lactation goals
* resides outside of Wisconsin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Successful Development of a Remote Collection Protocol reported as the final Reagent:Sample ratio | through study completion, anticipated to be 1 year
  The primary endpoint is generation of a remote collection protocol for use with a leading reagent in RNA preservation of human milk. There is no statistical test or null hypothesis associated with this endpoint, rather, a summary of relevant findings from all study secondary and exploratory endpoints.

SECONDARY OUTCOMES:
Concentration of RNA in Human Milk | through study completion, anticipated to be 1 year
  The concentration of extracted RNA (ng/uL) will be measured by a Qubit Fluorometer.
Purity of RNA in Human Milk | through study completion, anticipated to be 1 year
  The purity of extracted RNA will be measured by a Qubit Fluorometer. Purity will be assessed using wavelengths, the ratio of absorbance for A260/280 and A230/280.
RNA Integrity Number (RIN) | through study completion, anticipated to be 1 year
  Integrity of the extracted RNA will be measured using an agilent bioanalyzer. RIN is reported on a scale of 1 to 10 where higher numbers indicate higher integrity.
Quantitative PCR (qPCR) | through study completion, anticipated to be 1 year
  The epithelial cell and microRNA population will be quantified by measuring expression of epithelial cell and microRNA target genes.
Sample Collection Feasibility Data | data collected at time of sample return from participant (one time point greater than one month after lactation begins and within 7 days of sample collection)
  Participants answer 8-items scored on a 1 (discourage) to 10 (encourage) scale regarding participation in lactation research to assess factors that would facilitate their participation (use of own breast pump, ability to use breast pump, opportunity to privately express a sample in a clinic or at home, handling reagents with gloves, opportunity to participate in maternal and infant health research, opportunity to participate in genetic research).

OTHER OUTCOMES:
Perceived Stress Scale | data collected at time of sample return from participant (one time point greater than one month after lactation begins and within 7 days of sample collection)
  scored from 0-40 with higher scores indicating higher stress
Generalized Anxiety Disorder (GAD-7) | data collected at time of sample return from participant (one time point greater than one month after lactation begins and within 7 days of sample collection)
  Scores range from 0 to 21, with higher scores indicating greater anxiety.
Edinburgh Postpartum Depression Scale (EPDS) | data collected at time of sample return from participant (one time point greater than one month after lactation begins and within 7 days of sample collection)
  scored from 0-30 with higher scores indicating higher depression
MEDQ-Sus Questionnaire | data collected at time of sample return from participant (one time point greater than one month after lactation begins and within 7 days of sample collection)
  scored from 0-16 with higher scores indicating greater adherence to a Mediterranean dietary pattern

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Desorcy-Scherer, PhD, RN, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF